CLINICAL TRIAL: NCT00116974
Title: Periodontal Infection and Prematurity Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Protocol Expired. Terminated by IRB
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 801404
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Periodontal Diseases; Premature Birth
Keywords: Dental scaling
MeSH Terms: conditions — Periodontal Diseases; Premature Birth | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: Scaling and root planing
- 2 (Placebo Comparator)
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Procedure: Scaling and root planing — Scaling and root planing

SUMMARY:
This research project is a multi-center double-blind, parallel, randomized, controlled clinical trial design comparing the efficacy of dental scaling and root planing to control treatment (superficial cleaning) for the prevention of preterm birth in pregnant women with periodontal disease.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 6 and 20 completed weeks

Exclusion Criteria:

* Periodontal treatment during the pregnancy
* Antibiotic use within 2 weeks of enrollment
* Use of antimicrobial mouthwash within 2 weeks
* Multiple gestation
* Known mitral valve prolapse

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2004-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Whether screening and treating periodontal disease using scaling and root planing early in pregnancy can reduce the incidence of spontaneous preterm birth <35 weeks | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: George A Macones, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Jeffcoat M, Parry S, Sammel M, Clothier B, Catlin A, Macones G. Periodontal infection and preterm birth: successful periodontal therapy reduces the risk of preterm birth. BJOG. 2011 Jan;118(2):250-6. doi: 10.1111/j.1471-0528.2010.02713.x. Epub 2010 Sep 14. PMID 20840689